CLINICAL TRIAL: NCT00453804
Title: Injectable Versus Oral Naltrexone Treatment of Alcohol Dependence In Serious Mental Illness (SMI): A Pilot Study
Brief Title: Injectable Versus Oral Naltrexone Treatment of Alcohol Dependence In Serious Mental Illness (SMI)
Acronym: vivitrol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: Cephalon (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUNY UMU IRB # 5371
Record Dates: First submitted 2007-03-27; First posted 2007-03-29 (Estimated); Last update posted 2008-03-18 (Estimated); Status verified 2008-03

CONDITIONS: Bipolar Disorders; Schizophrenia; Schizoaffective Disorders; Alcohol Dependence
Keywords: Alcohol dependence; Major Mental Illness; Injectable naltrexone
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia; Psychotic Disorders; Alcoholism | interventions — Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: injectable naltrexone
Drug: oral naltrexone

SUMMARY:
The primary aim of this study is to determine the feasibility of long-acting injectable naltrexone administration in a clinical trial in patients with SMI who also have a diagnosis of alcohol dependence. Secondary aims include providing a preliminary assessment of the tolerability and safety of long-acting injectable naltrexone as compared with oral naltrexone in patients with SMI who also have a diagnosis of alcohol dependence. An additional aim is to provide a preliminary assessment of the efficacy of long-acting injectable naltrexone as compared with oral naltrexone in reducing alcohol use from baseline levels

DETAILED DESCRIPTION:
The overall goal of this project is to improve the treatment of alcohol abuse and dependence in patients with serious mental illness (SMI). SMI for this study is defined as any patient with any of the following diagnoses: schizophrenia, schizoaffective disorder, bipolar type I disorder, major depressive disorder with psychotic features, or psychotic disorder not otherwise specified. Alcohol and other substance use disorders (SUDs) are common among individuals with SMI such as schizophrenia. SUD comorbidity is associated with many adverse consequences. However, to date, few reports have addressed the efficacy of pharmacological treatments for SUDs in this population. Naltrexone pharmacotherapy is an effective treatment for alcohol dependence, but it has not been systematically applied to the care of patients with SMI. This pilot study plans to use a new intramuscular long-acting form of naltrexone that needs to be administered every 4 weeks compared to daily oral naltrexone, which we are also studying in this pilot. This could improve adherence to a medication regimen, which has been shown to be critical to successful naltrexone treatment of alcohol dependence. The proposed project is a 1-year pilot program of research. It is a randomized prospective parallel groups open-label trial of long-acting intramuscular (IM) naltrexone injected every 4 weeks compared to monthly prescriptions of oral naltrexone in a cohort of 20 subjects, ten for each treatment modality. The study is 16 weeks in duration, consisting of a 12-week course of naltrexone plus one follow-up interview at 4 weeks after discontinuation of medication. Voucher-based incentives are provided to all subjects to ensure attendance for medication administration. Weekly motivational counseling sessions are conducted and focus on improving motivation to stop alcohol use. Study outcomes consist of self-report and biological measures of alcohol use as well as measures of psychiatric symptom severity.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, age 18 to 69, with a DSM-IV diagnosis of Schizophrenia, Schizoaffective Disorder, Major Depressive Disorder (MDD) with Psychotic features, Bipolar Type I or Type II Disorder, or Psychosis not Otherwise Specified (NOS) Disorder;
2. DSM-IV diagnosis of Alcohol Dependence;
3. Level of Drinking:

   1. At least four days of drinking in the 30 days prior to consent and/or during screening period OR
   2. For prospective subjects who are currently in an inpatient or residential facility or recently discharged within 30 days prior to consent: At least 4 days of drinking during the period of time immediately prior to inpatient admission and/or during post-discharge.
4. Currently prescribed antipsychotic medications, mood stabilizers, or antidepressants.
5. One negative urine screen for opiates prior to start of medication and a self-report of no opioid use for at least 1 week prior to starting medication.
6. Currently involved in outpatient psychiatric treatment at one of the study sites (Hutchings Psychiatric Center, SUNY Upstate Adult Psychiatric Clinic, St. Joseph's Hospital, VA Medical Center) or at another location in the community.

Exclusion Criteria:

1. Inability to give adequate informed consent;
2. Currently taking disulfiram (Antabuse), naltrexone, or acamprosate (Campral);
3. Current DSM-IV diagnosis of Opioid Dependence;
4. Current regular use of prescribed opioid analgesics, such as methadone, morphine, codeine, meperidine, and all other opioids. If the subject reports taking a prescribed opioid analgesic only occasionally, the study physician or nurse practitioner will contact the prescribing physician regarding the safety of study participation and the possibility of using an alternative. The principal investigator will make the final determination after obtaining the primary physician's recommendation regarding this criterion.
5. Current daily use of non-prescribed opioids.
6. Currently taking ibuprofen or other potentially hepatotoxic medications in amount and/or frequency judged by the Principal Investigator to pose clinically significant added risk of hepatic injury;
7. Female patients of childbearing potential who are sexually active, not sterile, and who deny using birth control;
8. Female patients who are pregnant or nursing;
9. Significant unstable medical problems, including any significant unstable psychiatric disorders. The study physician conducting the medical history and physical exam will exclude such clinically unstable individuals;
10. AST (aspartate aminotransferase test) levels: If AST is greater than 3x upper limit of normal;
11. Subjects who do not attend required screening appointments. Subsequent exclusion from the study for reasons related to non-attendance will be based on the judgment of the principal investigator;
12. In need of acute medical detoxification from alcohol in the judgment of the study physician based on results a score of 12 or more on the Clinical Institute Withdrawal Assessment of Alcohol Scale Based on DSM-III-R (CIWA-AD) and other information obtained;
13. Scheduled surgery within 3 months of intake;
14. Subjects who have pending legal proceedings whose outcome may lead to incarceration within 3 months

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2006-07; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Primary: Measures of Alcohol Use; Psychiatric Symptom Severity

SECONDARY OUTCOMES:
adherence to medication, alcohol-related problems, quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Steven L Batki, MD, Principal Investigator — SUNY Upstate Medical University, Psychiatry Department
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

REFERENCES:
- [Result] Batki, S.L., Dimmock, J.A., Cavallerano, M., Leontieva, L., DeRycke, S., Ploutz-Snyder, R., Gallinger, L., Strutynski, K., Canfield, K., Carey, K.B., Maisto, S.A., Keegan, P., McMaster, T. (under review) (poster presentation) A pilot trial of oral versus long-acting injectable naltrexone in serious mental illness. Research Society on Alcoholism, 30th Annual Scientific Meeting 2007
- See also: SUNY Upstate Medical University — http://www.upstate.edu/